CLINICAL TRIAL: NCT03184948
Title: Understanding Neonatal Jaundice in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Merced (Other)
Collaborators: Rwanda Pediatric Association (Unknown); Ministry of Health, Rwanda (Other Government); Rwanda Bio-Medical Center (Unknown); Child Relief International (Unknown); D-Rev (Unknown)
Responsible Party: Principal Investigator, Ketki Sheth, Assistant Professor, University of California, Merced
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: FWA Assurance No: 00001973
Record Dates: First submitted 2017-06-05; First posted 2017-06-14 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Jaundice, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Intervention Model Description: Hospitals (i.e., participants) receive the intervention (i.e., Brilliance phototherapy device) at different times in the study. In the first phase, a set of hospital facilities receive the device. After three months of using the device, another set of hospital facilities receive the device. And after an additional three months (approximately 6 months after the first set of hospitals implemented their device), all hospitals will have been provided with the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 (Active Comparator): This is the first set of randomly selected hospitals to receive the intervention (Brilliance device). The intervention to be provided is the phototherapy device, Brilliance.
  *No individual participants are recruited for this study.
  Interventions: Device: Brilliance
- Phase 2 (Active Comparator): This is the second set of hospitals to receive the device. For the first three months, they receive no intervention, after which they become part of the "active comparator" arm. The intervention to be provided is the phototherapy device, Brilliance.
  *No individual participants are recruited for this study.
  Interventions: Device: Brilliance
- Phase 3 (No Intervention): This is the last set of hospitals to receive the device. For the first six months, they receive no intervention, after which the study is completed and they are given the device Brilliance.
  *No individual participants are recruited for this study.

INTERVENTIONS:
Device: Brilliance — The intervention is the provision of the Brilliance phototherapy machines to hospitals. This device is to be provided to facilities regardless of the study -- the study's involvement has been to collaborate with the Ministry of Health so that Brilliance is distributed in a randomized staggered method. In that sense, the study may be considered observational, as the study is not driving whether or not a hospital receives Brilliance, only when it receives Brilliance in a short time frame.
  Arms: Phase 1; Phase 2

SUMMARY:
This study exploits the distribution of low-cost high-quality phototherapy devices (Brilliance by D-Rev) to public hospitals in Rwanda to assess whether the provision of improved technology improves health care for infant jaundice. Specifically, the investigators are interested in measuring whether the provision of an additional high-quality phototherapy device, a known effective treatment for jaundice, successfully translates into improved care of neonatal jaundice in Rwanda where the burden of jaundice is particularly high.

DETAILED DESCRIPTION:
The Ministry of Health (MIH) in Rwanda has planned to provide Brilliance devices (phototherapy) to 46 public hospitals in Rwanda. The investigators have worked with MIH to have the delivery of these machines be staggered over three phases through random selection. The methodology relies on the staggered distribution of Brilliance devices and survey data collected prior and during delivery dates to evaluate the provision of low-cost high quality phototherapy machines, following the basic design of a staggered randomized controlled trial. Specifically, the investigators will survey all hospitals prior to the receipt of any Brilliance devices to provide a baseline description of the care received in these facilities. These surveys will collect information on the facility itself, including average infant jaundice caseloads and descriptions of recent cases. The investigators will then randomly select 15 hospitals to receive the Brilliance units. Three months after installation of Brilliance has occurred at these facilities (Group 1), another randomly selected subset of 16 facilities (Group 2) will receive their Brilliance machines. Three months after these installations have been completed, the remaining facilities (Group 3) will receive their Brilliance machines. During this period, there will be ongoing data collection from the hospitals, creating a panel dataset on the jaundice-related caseloads at these facilities. The data collected will be akin to collecting hospital records of patients diagnosed with jaundice, but no identifiable patient information will be collected.

ELIGIBILITY:
Inclusion Criteria:

* For patient level record (de-identified), diagnosed by the facility for having infant jaundice
* The facilities are included based on selection by the Ministry of Health for receiving additional phototherapy machines.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Length of treatment for infant jaundice | Through study completion, an average of 9 months
  Number of hours infant diagnosed with jaundice is provided phototherapy (PT). This is calculated by subtracting the age at which the patient is first given PT from the age at which the patient is removed from PT. The analysis is conditional on the subset of infants diagnosed with jaundice.
Length of hospital duration for infant jaundice | Through study completion, an average of 9 months
  This is measured by the duration of stay at the facility, as measured by the time between being admitted and being discharged. The analysis is conditional on the subset of infants diagnosed with jaundice.

SECONDARY OUTCOMES:
Increased rate of reduction in bilirubin | Through study completion, an average of 9 months
  Using different measures of estimated bilirubin levels for one patient and the age at which those tests were provided, we will estimate the change in bilirubin levels over the change in age (by hours) as the rate of reduction in bilirubin levels. This assumes that age at diagnosis is similar across treatment arms. If this is not the case or if our estimates are not precise, we will use maximum bilirubin levels recorded as a proxy. The analysis is conditional on the subset of infants diagnosed with jaundice.
Improved Treatment of Jaundice | Through study completion, an average of 9 months
  An indicator variable for whether the patient was treated at the facility (as opposed to being referred elsewhere for treatment).
Improved Treatment of Jaundice By Not Being Referred Elsewhere | Through study completion, an average of 9 months
  An indicator variable for whether the patient was treated at the facility (as opposed to being referred elsewhere for treatment).
Improved Treatment of Jaundice by Receiving Phototherapy | Through study completion, an average of 9 months
  An indicator variable for whether the patient received phototherapy.
Improved Treatment of Jaundice by Not Sharing Phototherapy | Through study completion, an average of 9 months
  An indicator variable for whether the patient did not share a phototherapy machine with another infant
Improved Treatment of Jaundice by Using Single Phototherapy Device | Through study completion, an average of 9 months
  An indicator variable for whether the patient used multiple phototherapy machines;
Improved Treatment of Jaundice by Reducing Exchange Transfusions | Through study completion, an average of 9 months
  An indicator variable for whether the patient received an exchange transfusion
Improved Treatment of Jaundice by Not Meeting Threshold for Exchange Transfusion | Through study completion, an average of 9 months
  An indicator variable for whether the patient reached the threshold for exchange transfusion

OTHER OUTCOMES:
Age at time of jaundice diagnosis | Through study completion, an average of 9 months
  Average age of infant at the time of jaundice diagnosis
Jaundice diagnosis rates | Through study completion, an average of 9 months
  Rate of infant jaundice diagnoses per month per admitted infants as reported by hospital facility
Jaundice diagnosis levels | Through study completion, an average of 9 months
  Number of infant jaundice diagnoses per month as reported by the hospital facility
Fee Charged | Through study completion, an average of 9 months
  Reduction in cost of jaundice case (fee charged and amount earned by facility per diagnosed jaundice patient) as reported by hospital facility.
Increased technical capacity by Number of Phototherapy Devices | Through study completion, an average of 9 months
  Number of Phototherapy machines at facility
Increased technical capacity by Number of Operational Phototherapy Devices | Through study completion, an average of 9 months
  Number of operational phototherapy machines at facility
Increased technical capacity by Improved Irradiance Levels | Through study completion, an average of 9 months
  Average irradiance levels of phototherapy machines at the hospital facility

CONTACTS AND LOCATIONS:
Overall Officials: Ketki Sheth, PhD, Principal Investigator — University of California, Merced; Lisine Tuysenge, MD, Principal Investigator — Rwanda Pediatric Association
Locations (1):
- University Central Hospital of Kigali, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Undecided
All IPD collected will be anonymized and aggregated for analysis. The anonymized information will be shared publicly if permission from the Rwandan Ministry of Health is granted.

REFERENCES:
- Available data/document: Statistical Analysis Plan — http://ketkisheth.weebly.com/